CLINICAL TRIAL: NCT03161015
Title: A Non-Randomized, Open-Label, Parallel Group, Single-Dose Study to Compare the Pharmacokinetics of GBT440 in Subjects With Renal Impaired Function to Healthy Subjects
Brief Title: Single-Dose PK Study of GBT440 in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GBT440-0110
Record Dates: First submitted 2017-05-08; First posted 2017-05-19 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — voxelotor

STUDY DESIGN:
Intervention Model Description: Multiple-center, nonrandomized, open-label, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GBT440 Dose 1: Severe Renal Impairment (Experimental): eGFR < 30 mL/min/1.73m2, not on dialysis
  Interventions: Drug: GBT440
- GBT440 Dose 1: Moderate Renal Impairment (Experimental): 30 mL/min/1.73m2 = or < eGFR < 60 mL/min/1.73m2
  Interventions: Drug: GBT440
- GBT440 Dose 1: Mild Renal Impairment (Experimental): 60 mL/min/1.73m2 = or < eGFR < 90 mL/min/1.73m2
  Interventions: Drug: GBT440
- GBT440 Dose 1: Normal Renal function (Experimental): eGFR > or = 90 mL/min/1.73m2
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — Oral

SUMMARY:
A Phase 1, multiple center, nonrandomized, open-label, parallel group study of a single oral dose of GBT440 administered in subjects with mild, moderate, or severe renal impairment disease and healthy subjects with normal renal function.

DETAILED DESCRIPTION:
Up to 40 adult subjects will be enrolled. Safety and PK assessments will be performed at selected time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Males or females, 18 to 80 years old
* Willing and able to give written informed consent

Subjects with renal impairment:

* Severe renal impairment (eGFR < 30 mL/min/1.73m2, not on dialysis)
* Moderate renal impairment (30 mL/min/1.73m2 = or < eGFR < 60 mL/min/1.73m2)
* Mild renal impairment (60 mL/min/1.73m2 = or < eGFR < 90 mL/min/1.73m2)

Healthy subjects:

* Match in age, gender and body mass index with renal impaired subjects
* Healthy and without clinically significant abnormalities in vital signs, ECGs, physical exam, clinical laboratory evaluations, medical and surgical history

Exclusion Criteria:

All subjects:

* Participation in another clinical trial of an investigational drug (or medical device) within 30 days of the last dose of investigational drug or 5 half lives whichever is longer, prior to screening, or is currently participating in another trial of an investigational drug (or medical device)
* Any signs or symptoms of acute illness at screening or Day -1
* History or presence of clinically significant allergic, hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease

Subjects with renal impairment:

- History of clinically significant hepatic disease e.g. hepatitis, cirrhosis and or liver enzymes (ALT, AST, GGT and total bilirubin) > 5 times the upper limit of normal within the past year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Cmax of GBT440 in subjects with severe, moderate, or mild renal impairment versus subjects with normal renal function | 28 days max
  Maximum observed plasma concentration
Tmax of GBT440 in subjects with severe, moderate, or mild renal impairment versus subjects with normal renal function | 28 days max
AUC of GBT440 in subjects with severe, moderate, or mild renal impairment versus subjects with normal renal function | 28 days max
T1/2 of GBT440 in subjects with severe, moderate, or mild renal impairment versus subjects with normal renal function | 28 days max

SECONDARY OUTCOMES:
Number of subjects with treatment-related Adverse events | 28 days max

CONTACTS AND LOCATIONS:
Overall Officials: Carla Washington, Study Director — Global Blood Therapeutics
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - OCRC, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided